CLINICAL TRIAL: NCT07358377
Title: An Open-Label, Multi-Center Phase II Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of HRS-6209 in Combination With Fulvestrant or Letrozole in Patients With Solid Tumor
Brief Title: To Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HRS-6209 in Subjects With HR-Positive/HER2-Negative Solid Tumor
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-6209-205
Record Dates: First submitted 2025-12-28; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HRS-6209 Capsules and fulvestrant injection (Experimental)
  Interventions: Drug: HRS-6209 Capsules and fulvestrant injection

INTERVENTIONS:
Drug: HRS-6209 Capsules and fulvestrant injection — HRS-6209, 100mg BID for 4 weeks, and single dose of fulvestrant injection

SUMMARY:
To evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HRS-6209 in Subjects with HR-Positive/HER2-Negative solid tumor.

ELIGIBILITY:
Inclusion Criteria

1. Ability to understand the trial procedures and possible adverse events, voluntarily participate in the trial.
2. Adequate bone marrow and other vital organ functions
3. Adequate liver function tests
4. HR-positive or HER2-negative solid tumor patients

Exclusion Criteria

1. Plan to receive any other anti-tumor therapy during the study.
2. Active brain metastases .
3. Have poorly controlled or severe cardiovascular disease, including (1) congestive heart failure.
4. Previous use of fulvestrant
5. clinically significant endometrial abnormalities, including but not limited to endometrial hyperplasia and dysfunctional uterine bleeding.
6. With uncontrollable chronic systemic complications (such as severe chronic lung, liver, kidney, or heart disease).
7. With acute or active tuberculosis infection requiring medication.
8. Pregnant or lactating women, or females planning to become pregnant During the study.
9. Known history of clinically significant liver disease, untreated active hepatitis (hepatitis B, defined as hepatitis B virus surface antigen [HBsAg] or hepatitis B core antibody [HBcAb] positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-04-10 (Estimated); Study Completion 2027-11-10 (Estimated)

PRIMARY OUTCOMES:
Safety by reporting incidence and severity of Adverse events (graded as per CTCAE V5.0) of adverse events (AEs) and serious adverse events (SAEs), | Screening up to study completion,, an average of 1 year.
  To safety and tolerability of HRS-6209 in combination with fulvestrant in patients with advanced unresectable or metastatic breast cancer

SECONDARY OUTCOMES:
Concentration | From administration to C2, up to 4 months.
  Plasma concentrations of HRS-6209 during multiple dosing, directly observed from data.
Cmax,ss | From administration to C2, up to 4 months.
  Css, max are steady-state maximum concentrations of HRS-6209 during multiple dosing, and are directly observed from data.
Cmin,ss | From administration to C2, up to 4 months.
  Css, min are the steady-state trough concentrations of HRS-6209 during multiple dosing, and are directly observed from data.
Objective Response Rate (ORR) | Screening up to study completion, an average of 2 years.
  ORR refers to the proportion of subjects with a complete response (CR) or partial response (PR) based on all soft tissue assessments recorded from the date of first drug administration to either the date of radiographic disease progression (including bone progression and soft tissue progression), death from any cause, or the initiation of a new antitumor therapy, whichever occurs first. For subjects with CR or PR at the first evaluation, the efficacy should be confirmed 4 weeks later or at the next tumor imaging evaluation. The numerator includes subjects with a confirmed CR/PR at least 4 weeks after the initial assessment. The denominator consists of subjects with measurable target lesions at baseline.
Best of Response (DoR) | Screening up to study completion, an average of 2 years.
  BOR refers to the best response of tumor evaluation, including CR, PR, stable disease (SD), progressive disease (PD), and not evaluable for response (NE).
Disease Control Rate (DCR) | Screening up to study completion, an average of 2 years.
  DCR refers to the time from the first occurrence of CR or PR to PD or death from any cause, whichever occurs first, in subjects with objective response. DCR will be recorded from baseline visit until the end of the study.
rPFS (radiographic progression-free survival | Screening up to study completion, an average of 2 years.
  rPFS refers to the time from the first dose of investigational drug to the first radiographic PD or death from any cause (whichever occurs first) as assessed by the investigator. rPFS will be recorded from baseline visit until the end of the study.